CLINICAL TRIAL: NCT00408473
Title: A Randomised Double-blind Pilot Study Comparing Flecainide CR and Placebo in the Early Treatment of Patients With a Documented First Episode of Atrial Fibrillation.
Brief Title: Comparative Study of Flecainide CR and Placebo in the Early Treatment of Atrial Fibrillation.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: 3M (Industry)
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1556-FLEC
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2007-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Flecainide

INTERVENTIONS:
Drug: Flecainide

SUMMARY:
The purpose of the study is to assess the efficacy of flecainide controlled release (CR) in the prevention of recurrent AF during 9 months of active treatment compared to placebo in patients with only one documented AF episode.

ELIGIBILITY:
Inclusion Criteria:

* History of first symptomatic & documented episode of AF
* LVEF > 40% and not on AAD and in sinus rhythm at time of recruitment

Exclusion Criteria:

* History of more than 1 symptomatic documented AF episode, persistent or permanent AF.
* History of ablation for previous AF
* Reversible cause for AF (e.g.thyroid, alcohol, pulmonary embolism, surgery
* Severe symptoms during AF episode (e.g.syncope, chest pain)
* All types of treated arrhythmias other than AF
* History of myocardial infarction (MI), coronary artery disease (CAD), heart failure (I, II, III and IV of New York Heart Association -NYHA- classification) or valvular diseases
* Left ventricular ejection fraction (LVEF) ≤ 40%
* Bradycardia < 40 beats/min and all ECG abnormalities: PR> 240ms or QRS> 120 ms or QTc> 440 ms
* Brugada syndrome
* Conduction disturbances: complete bundle branch block (LBBB) or (RBBB), bifascicular block
* 2nd or 3rd degree atrioventricular (AV) block
* Sinus node dysfunction
* Severe hypertension with:Systolic blood pressure ≥ 180 mmHg, and / or· Diastolic blood pressure ≥ 100 mmHg
* Left ventricular hypertrophy (LVH) with septal thickness > 14 mm on Echocardiogram
* Implanted pacemaker
* Heart surgery within the last 6 months, or non-stable postoperative condition
* Renal failure: serum creatinine ≥ 150 µmol/l or creatinine clearance ≤ 50 ml/min (Cockroft and Gault formula
* Uncorrected electrolytic abnormalities
* Have used recently in the last 3 months prior to the inclusion any of the following treatments: Oral amiodarone, Treatments that lengthen QT interval (e.g.Sultopride, Drugs causing torsades de pointe (e.g.mizolastine, pentamidine, sparfloxacin, moxifloxacin, Bupropion
* Anti-hypertensive drugs other than permitted in the study: ACE-I, ARB (sartans) and DHP from Calcium channel blockers (CCB

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256

PRIMARY OUTCOMES:
Time to the first relapse after randomization, with or without symptoms documented on ECG, Holter or "Self ECG unit" recording.

SECONDARY OUTCOMES:
Total number of AF recurrences during the treatment period
Total number of patients in sinus rhythm at the end of the study
AF Burden
Number of emergency admissions due to AF recurrence
Cardiac Safety

CONTACTS AND LOCATIONS:
Overall Officials: Prof E Aliot, Principal Investigator — CHU Brabois, avenue de Bourgogne, 54511 Vandoeuvre-les-Nancy. FRANCE
Locations (47):
- Belgium (5):
  - Imeldaziekenhuis, Imeldalaan 9, Bonheiden
  - Hôpital St.-Joseph, Rue de la Duchère 6, Gilly
  - Virga Jesse Ziekenhuis, Stadsomvaart 11, Hassel
  - Regionaal Ziekenhuis Heilig Hart, Naamsestraat 105, Leuven
  - Clinique Sainte-Elisabet, Place Louise Godin 1, Namur
- Bulgaria (10):
  - Department of Cardiology, MHAT Burgas AD, 73 Stefan Stambolov blvd, Burgas
  - Cardiology Clinic and ICU, UMHAT "Dr. Georgi Stranski" EAD, 8a Georgi Kochev Str, Pleven
  - Intensive Therapeutic Department, MHAT Ruse, 2 Nezavosimost str, Rousse
  - Clinic of cardiology at Second MHAT, 120, Hristo Botev Blvd, Sofia
  - National Cardiology Hospital EAD, 65 Konjovitza Str., Sofia
  - Department of Internal medicine II, University hospital "Aleksandrovska" , 1 G. Sofiyski str, Sofia
  - Clinic of Cardiology, University Hospital 'Queen Giovanna', 8 Bialo More str, Sofia
  - Department of Emergency and Intensive care, Military Medical Academy, 3 G. Sofiisky str, Sofia
  - Intensive care unit - MHATEM "Pirogov" , 21 Totleben Blvd, Sofia
  - CCU, University Hospital "St. Marina" , 1 Hristo Smirnenski Blvd, Varna
- France (18):
  - Centre Hospitalier Général, 22, boulevard Général Sibille, Albi
  - Hôpital d'Arras service de cardiologie, 57 avenue Wiston Churchill, Arras
  - Philippe CHEMIN, 49 rue du Bocage, Bordeaux
  - Hopital d'instruction des armées, rue Colonel Fonferrier, Brest
  - Centre Hospitalier Général, 516 avenue de Paris, Cambrai
  - Patrick GIRAUD, Bat C 132 av Gabriel Péri, Cavaillon
  - André CORBIN, 28 rue du Conte de la Garaye, Dinan
  - Centre Hospitalier du Leman, 3 avenue de la dame, Evian-thonon
  - Verschuersen Iordanka, 4 rue Béranger, Fontainebleau
  - Hôpital de Freyming Merlebach- Service de Cardiologie, 2 rue de France, Freyming-Merlebach
  - Centre Hospitalier Général, 10 rue de la Charité, Langres
  - Jean Claude GICHTENAERE, 8 quai du Général Leclerc, Martigues
  - CHI Montfermeil, 10 rue du Gal Leclerc, Montfermeil
  - Résidence Médicale Les Roses, 57, route de Lavérune, Montpellier
  - Patrick KOHAN, 18 rue de la Commanderie, Nancy
  - Centre Hospitalier Regional, 1 rue du Friscaty, Thionville
  - Hôpital d'Instruction des Armées Sainte Anne, Boulevard Sainte Anne, Toulon
  - Centre médical, Promenade du petit Languedoc, Villefranche-de-Rouergue
- Germany (6):
  - Zentralklinic Bad Berka Gmbr Klinic fur Kardiologie- Leitender Arzt der Avteilung - Rhythmologie und invasive Elektrophysiologie, Robert Koch Allee 9, Bad Berka
  - Director of Electrophysiology Laboratory - Department of Medicine - Cardiology- University of Bonn, Sigmund Freud Str 25 -, Bonn
  - Klinikum Coburg , Ketschendorfer Str. 33, Coburg
  - Div Cardiology; University Hospital , Leipzigen St 44 -, Magdeburg
  - Oberarzt Medizinische Klinik und Poliklinik C IZKF Münster Kompetenznetzt Vorhofflimmern Universitätsklinikum Münster, Albert-Schweitzer-Straße 33,, Münster
  - Kardiologische Praxis, Magirusstr.49, Ulm
- "Academisch Ziekenhuis Maastricht, P. Debyelaan 25, Maastricht, Netherlands
- Romania (6):
  - SPITALUL JUDETEAN-SECTIA CARDIOLOGIE, BRASOV, Str. Independentei Nr. 1, Brasov
  - "SPITALUL CLINIC DE URGENTA ""ELIAS""-Clinica de Cardiologie, Str. Marasti, Nr. 17, sect 1, Bucharest
  - Spitalul Clinic Colentina-Departamentul Cardiologie, str. Stefan cel Mare, nr. 19-21, sector 2, Bucharest
  - "SPITALUL CLINIC de RECUPERARE, Str. Viilor Nr.46-50, Cluj-Napoca
  - Centrul de Cardiologie , Str. Tabaci No. 1, Craiova
  - CARDIO EXPERT, Str. Romulus, Nr. 62., Timișoara
- Hospital Universitario de Getafe, Carretera de toledo, Madrid, Spain